CLINICAL TRIAL: NCT02488941
Title: Mapping of Metabolic Liver Functions in Patients With Non-alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Metabolic liver function NAFLD
Record Dates: First submitted 2015-06-17; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Liver Function Tests; Blood Coagulation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy Blood : serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Non-alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in the western world and an important cause of morbidity and mortality including risk of cardiovascular disease. A ruling dogma is that a fatty liver is well-functioning. Recent studies imply the contrary but quantitative measurements of metabolic liver function have not been systematically investigated in NAFLD.

Objectives: To study and quantify specific metabolic liver functions in varying degrees of NAFLD. Furthermore to map the coagulation system of patients with NAFLD.

Methods: A human clinical study. Metabolic liver functions are studied by a series of functional tests (Galactose elimination capacity (GEC), Aminopyrine breath test (ABT), Indocyanine green plasma disappearance rate (ICG-PDR), Functional hepatic nitrogen clearance (FHNC)). Regional liver function evaluated by 2-[18F]fluoro-2-deoxy-D-galactose (FDGal) PET/CT is compared to fat infiltration assessed by Magnetic resonance imaging (MRI). Primary and secondary hemostasis, natural anti-coagulants and fibrinolysis are evaluated.

Perspectives: To challenge the dogma, that hepatic metabolic function is not affected in NAFLD, improving the understanding of the relationship between the clinical degree of NAFLD, histology, metabolic functions, and imaging. Furthermore to disclose a proposed procoagulant imbalance in NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Hepatic steatosis found on ultrasound
* Clinical indication for liver biopsy (typically persistently elevated alanine transaminase (ALT) levels)

Exclusion Criteria:

* Other liver pathology
* Alcohol consumption > 20g/day
* Chronic inflammatory disease, current infection or cancer
* Diabetes mellitus type I, II or HbA1c ≥ 48 mmol/mol (6.5 %)
* Prednisolone treatment within last 8 weeks
* Pregnancy within last 12 months
* Contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with varying degrees of NAFLD
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Metabolic Liver Function assessed by GEC | Baseline
Metabolic Liver Function assessed by FHNC | Baseline
Metabolic Liver Function assessed by ABT | Baseline
Metabolic Liver Function assessed by ICG-PDR | Baseline
Regional metabolic liver function evaluated by FDGal PET/CT | Baseline
  100 megabecquerel FDGal is injected intravenously in the beginning of a 20 min PET recording and 3D images of regional metabolic liver function expressed in terms of hepatic metabolic clearance of FDGal is created.
Regional fat infiltration assessed by MRI | Baseline

SECONDARY OUTCOMES:
Primary hemostasis | Baseline
Secondary hemostasis | Baseline
Natural anti-coagulants | Baseline
Fibrinolysis | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Professor, Study Director — Department of Hepatology & Gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology & Gastroenterology, Aarhus, Denmark